CLINICAL TRIAL: NCT04687865
Title: Biological Material Bank for Studies Related to Organ Transplantation
Brief Title: Constitution of a Biobank for Studies Related to Organ Transplantation (Lyon Centaure Biocollection)
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0964
Record Dates: First submitted 2020-12-16; First posted 2020-12-29 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Organ Transplantation
MeSH Terms: interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biobank — For each patient included in the study the following samples will be collected at the indicated time points after transplantation:
  * Serum samples and plasma sample: Day1, Month 1, Month 3, Month 6, Month 12, month 60, month 120 and at the time of each allograft biopsy.
  * Urines samples: Month 3 and Month 12 and at the time of each allograft biopsy.
  * Peripheral Blood Mononuclear Cell (PBMC): for each organ allograft biopsy.
  * Allograft biopsies: systematically at Month 3, and Month 12, and for cause in case of allograft dysfunction.

SUMMARY:
This study aims to constitute a collection of biological materials from in transplant patients and to provide biological materials from transplanted patients in order :

i) validate new theory on the cause of allograft loss, ii) develop innovative biomarker for rejection and other transplantation-related conditions (such as BK virus nephropathy, Post-transplant lymphoproliferative disorder ( PTLD) ...)

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patient ≥18 years old
* Recipient of an organ transplant
* Written informed consent

Exclusion Criteria:

* Non-affiliation to a social security system.
* Subjects deprived of liberties
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients that received a solid organ transplant at the transplantation department of Lyon University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2040-01-08 (Estimated); Study Completion 2040-01-08 (Estimated)

PRIMARY OUTCOMES:
the biological samples | At inclusion
  The goal of this study is to provide biological materials from transplanted patients
Change Biological Samples | Month 1
  The goal of this study is to provide biological materials from transplanted patients
Change Biological Samples | Month 3
  The goal of this study is to provide biological materials from transplanted patients
Change Biological Samples | Month 6
  The goal of this study is to provide biological materials from transplanted patients
Change Biological Samples | Month 12
  The goal of this study is to provide biological materials from transplanted patients
Change Biological Samples | Month 60
  The goal of this study is to provide biological materials from transplanted patients
Change Biological Samples | Month 120
  The goal of this study is to provide biological materials from transplanted patients

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Thaunat, MD, Principal Investigator — Edouard Herriot Hospital - Transplantation department
Locations (1):
- Hopital Edouard Herriot, Lyon, Rhône, France